CLINICAL TRIAL: NCT02789475
Title: DP-R212 Pharmacokinetic Study
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Alvogen Korea (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DP-CTR-212-I-01
Record Dates: First submitted 2016-05-23; First posted 2016-06-03 (Estimated); Last update posted 2016-06-03 (Estimated); Status verified 2016-05

CONDITIONS: Hypertension; Hyperlipidemias
MeSH Terms: conditions — Hypertension; Hyperlipidemias | interventions — Amlodipine; Rosuvastatin Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- amplodipine group (Experimental): Amlodipine for 8 days and Amlodipine+Rosuvastatin for 5 days
  Interventions: Drug: Amlodipine; Drug: Rosuvastatin
- rosuvastatin group (Experimental): Rosuvastatin for 5 days and Amlodipine+Rosuvastatin for 8 days
  Interventions: Drug: Amlodipine; Drug: Rosuvastatin

INTERVENTIONS:
Drug: Amlodipine — Amlodipine administration
Drug: Rosuvastatin — Rosuvastatin administration

SUMMARY:
An open-label, multiple-dose study to evaluate the pharmacokinetic drug-drug interaction of amlodipine and rosuvastatin in healthy adult male subjects.

ELIGIBILITY:
Inclusion Criteria:

* BMI 18-29
* signed the informed consent form prior to the study participation

Exclusion Criteria:

* Clinically significant disease
* Previously donate whole blood within 60 days or component blood within 14 days
* Clinically significant allergic disease
* Taken IP in other trial within 90 days
* An impossible one who participates in clinical trial by investigator's decision including laboratory test result

Ages: 19 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Estimated)
Dates: Start 2016-05; Primary Completion 2016-07 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
AUCτ,ss of Amlodipine and Rosuvastatin | 0,0.5,1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 24 hr
Cmax,ss of Amlodipine and Rosuvastatin | 0,0.5,1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 24 hr

CONTACTS AND LOCATIONS:
Overall Officials: Chul woo Kim, Ph.D., Principal Investigator — Inha University Hospital
Locations (1):
- Inha university hospital, Jung-gu, Incheon, South Korea

IPD SHARING:
Plan to Share IPD: No